CLINICAL TRIAL: NCT05190926
Title: Smart Technology for Anorexia Nervosa Recovery: A Pilot Intervention for the Post-Acute Treatment of Anorexia Nervosa
Brief Title: Smart Technology for Anorexia Nervosa Recovery
Acronym: STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other); Purdue University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00141926
Record Dates: First submitted 2021-12-08; First posted 2022-01-13 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Adolescents; Smartphone; Therapy Support Tools
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Treatment for Anorexia Nervosa Recovery (STAR) app (Experimental): STAR incorporates elements from the Unified Protocol and Acceptance and Commitment Therapy to reduce emotion avoidance and improve disordered-eating behaviors and negative emotions. Participants will complete 1-2 weekly modules in STAR for 12 weeks. During this time, participants will continue working with their outpatient therapist. Outcome and target engagement measures will be assessed daily or weekly within the STAR app. Participants will complete additional measures of outcome and target engagement at 3-months and 6-months after treatment. Parents will be asked to complete outcome measures at baseline, 12 weeks, 3-months, and 6-months.
  Interventions: Behavioral: Smart-Treatment for Anorexia Nervosa Recovery (STAR)
- Present-focused Anorexia Nervosa Coping Treatment (PACT) app (Placebo Comparator): PACT is an adapted form of Present-Centered Therapy and focuses on daily life stressors, problems, and concerns that may impact AN. Participants will complete 1 weekly module in Weeks 1, 2, and 12 and complete a Daily Diary of life stressors thereafter for 9 weeks. During this time, participants will continue working with their outpatient therapist. Outcome and target engagement measures will be assessed daily or weekly within the PACT app. Participants will complete additional measures of outcome and target engagement at 3-months and 6-months after treatment. Parents will be asked to complete outcome measures at baseline, 12 weeks, 3-months, and 6-months.
  Interventions: Behavioral: Present-focused Anorexia Nervosa Coping Treatment (PACT)

INTERVENTIONS:
Behavioral: Smart-Treatment for Anorexia Nervosa Recovery (STAR) — Adolescents will use their smartphone to access short 5-10 minute "modules" that teach them about the function of emotions, ways to regulate challenging emotions, and strategies to improve negative thinking, mood, and reduce eating-disorder symptoms. Module content will include text, images, videos, and interactive questions and quizzes.
  Arms: Smart Treatment for Anorexia Nervosa Recovery (STAR) app
Behavioral: Present-focused Anorexia Nervosa Coping Treatment (PACT) — Adolescents will use their smartphone to access two brief psychoeducational modules that teach about the common symptoms of AN, common reactions and problems associated with AN, and goals for treatment. Starting in Week 3, adolescents will complete a Daily Diary that will ask them to record life stressors, challenges, and problems, which will serve as a launching point for discussion with their outpatient therapist.
  Arms: Present-focused Anorexia Nervosa Coping Treatment (PACT) app

SUMMARY:
Anorexia nervosa (AN) has the highest mortality rate of any mental illness, with a typical onset in adolescence. Although family-based interventions are efficacious for up to 75 percent of adolescents with AN, approximately 30 percent will relapse after recovery. There is a critical need to improve treatments and prevent post-discharge relapse following acute treatment to improve outcomes for adolescents with AN.

To address this critical need, the investigators developed an adaptive smart-phone based therapy support tool for teens with AN, called Smart Treatment for Anorexia Recovery (STAR). STAR is for adolescents between the ages of 13-21 who recently received acute treatment for AN (e.g., inpatient, residential, intensive outpatient, or day hospital) who are currently working with an outpatient therapist. STAR incorporates elements from the Unified Protocol and Acceptance and Commitment Therapy to target emotion avoidance, which the investigators hypothesize will lead to reductions in eating-disorder behaviors. The investigators will compare STAR to Present-focused Anorexia Nervosa Coping Treatment (PACT), which focuses on current life stressors and problems.

The investigators' hypothesis is that STAR will improve outpatient treatment response and reduce relapse in adolescents discharged from intensive treatment for AN. The investigators will evaluate their hypotheses in two conditions: 1) STAR app and 2) PACT app. In both conditions, participants must be working with an individual outpatient therapist.

DETAILED DESCRIPTION:
AN is the third leading cause of chronic illness in adolescents and, if left untreated, can lead to major organ damage, structural and functional brain changes, and early-onset osteopenia and osteoporosis. Although family-based interventions are efficacious for up to 75% of adolescents with AN, approximately 30% will relapse after recovery. There is a critical need to optimize treatments and prevent post-discharge relapse following acute treatment to improve outcomes for adolescents with AN. To address this critical need, the investigative team developed a suite of digital tools that advance the science of assessment, risk prediction, and clinical-decision support for use in the post-acute treatment window, called "Smart Treatment for Anorexia Recovery (STAR)." STAR uses cutting-edge assessment technology to shorten test administration and machine-learning to predict likelihood of recovery. This information is then provided back to the clinician via an easy-to-use clinical-decision support tool to alert the clinician when user-entered data suggests the patient is not progressing.

In the current clinical trial, the investigators will expand STAR to test an adaptive mHealth intervention delivered in the post-discharge window. The investigators' hypothesis is that a transdiagnostic assessment and clinical-decision support tool delivered within the STAR suite will optimize face-to-face clinical service and the addition of an adaptive mobile-health (mHealth) intervention will improve outpatient treatment response and reduce relapse in adolescents discharged from intensive treatment for AN. The investigators' previous work supports the hypothesis. Specifically, the investigators' past studies provide robust support for the predictive validity and clinical utility of the investigators' assessment tool for predicting ED-related psychiatric impairment and recovery. However, the number of items across the paper-based assessment tool is 144, which is overly long for routine use. To overcome this challenge, the investigators developed a mobile phone app that uses computerized adaptive testing to reduce assessment length by up to 50% while retaining the reliability and validity of the original paper-and-pencil measure. The investigators propose to leverage this innovation to optimize both face-to-face and mHealth treatment for AN. The objectives are to: 1) develop the mHealth intervention (with clinician and stakeholder input) and 2) establish feasibility, acceptability, and preliminary effect size of the mHealth intervention using both clinician and patient data. To accomplish these objectives, the investigators will employ a computerized adaptive test coupled with machine learning algorithms, delivered within the app to signal clinicians when their clients are at-risk for poor outcomes and relapse. Specific aims include: 1) adapt the existing clinical tool to provide therapist support modules and patient mHealth messages; 2) conduct a preliminary randomized controlled trial (RCT) of the integrated assessment and mHealth intervention tool; 3) test preliminary mechanisms that lead to changes in AN symptoms.

STAR incorporates elements from the Unified Protocol and Acceptance and Commitment Therapy to target emotion avoidance, which the investigators hypothesize will lead to reductions in eating-disorder behaviors. The investigators will compare STAR to Present-focused Anorexia Nervosa Coping Treatment (PACT), which focuses on current life stressors and problems. The investigators' hypothesis is that STAR will improve outpatient treatment response and reduce relapse in adolescents discharged from intensive treatment for AN. The investigators will evaluate hypotheses in two conditions: 1) STAR app and 2) PACT app. In both conditions, participants must be working with an individual outpatient therapist.

Given there is a scarcity of specialty care for AN following acute treatment, yet 95% of adolescents have smartphones, the proposed research is innovative and significant because it has the future potential to reduce relapse and optimize existing community-delivered interventions for AN over the post-acute treatment window.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 21
* Able to read and speak fluent English
* Access to a smartphone
* Received acute treatment for anorexia nervosa or atypical anorexia nervosa [residential, inpatient, partial hospitalization (PHP), or intensive outpatient program (IOP)] within the past three months
* Currently receiving weekly outpatient treatment (or planning to start outpatient treatment) for current anorexia nervosa/atypical anorexia nervosa, or past anorexia nervosa/atypical anorexia nervosa (e.g., anorexia nervosa in partial remission).

Exclusion Criteria:

* Uncorrected visual impairments that would prevent smartphone use
* Intellectual or developmental disability
* Medical condition that affects appetite or weight (e.g., thyroid disorder, diabetes, cancer, pregnancy)
* Current psychotic disorder or substance use disorder
* BMI-z < 14 or lab abnormalities indicating medical instability
* Unwillingness for data to be shared with outpatient therapist

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index Z-Scores (BMI-z) | Baseline, 12-week intervention (weekly), and 3- and 6-month follow-ups
  Therapists, caregivers, or primary care physicians will provide weight and height measurements each week to calculate BMI-z.

SECONDARY OUTCOMES:
Change in Categorical Recovery Status | Baseline, 12-week, and 3- and 6-month follow-ups
  Responses from the Eating Disorder Diagnostic Survey (EDDS) will calculate categorical recovery status for anorexia nervosa (excellent, good, marginal, poor) based on definitions from Bardone-Cone et al. (2010). Baseline recovery status will allow the investigators to assess initial recovery status following acute treatment for anorexia nervosa.
Change in Mood and Anxiety Symptoms | Baseline, 12-week, and 3- and 6-month follow-ups
  The Mood and Anxiety Symptoms Questionnaire (MASQ) was designed to measure dimensions of mood and anxiety relevant to the Unified Protocol (General Distress, Anxiety, and Positive Affect). The investigators will use the MASQ to assess changes in internalizing symptoms over the course of treatment.
Change in Eating Disorder Symptom Severity | Baseline, 12-week, and 3- and 6-month follow-ups
  The investigators will use the total number of eating-disorder symptoms from the Eating Disorder Diagnostic Survey (EDDS) as an indicator of eating-disorder symptom severity.
Change in Psychiatric Impairment | Baseline, 12-week, and 3- and 6-month follow-ups
  Psychiatric and psychosocial impairment questionnaires will include the Clinical Impairment Assessment (CIA), which measures psychosocial impairment secondary to eating-disorder features and the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0).
Change in Parent-Reported Mealtime Behaviors | Baseline, 12-week, and 3- and 6-month follow-ups
  Parents will complete the Meals in Our Households (MOH) to measure: Structure of Family Meals; Parental Concern about Child's Diet; Spousal Stress Related to Mealtime Behaviors (if relevant); and Problematic Child Mealtime Behaviors.
Change in Emotion Avoidance | Baseline and 12-week intervention (weekly)
  The Brief Experiential Avoidance Questionnaire (BEAQ) will assess unwillingness to remain in contact with distressing emotions, thoughts, memories, and physical sensations. The investigators will use the BEAQ to test whether changes in emotion avoidance leads to changes in eating-disorder behaviors.
Change in Eating-Disorder Behaviors | Daily during the 12-week intervention period
  The investigators will use an ad-hoc checklist within the app to measure eating-disorder behaviors (e.g., binge eating, purging, etc.)
Change in Patient Skill Utilization | Daily during the 12-week intervention period
  Skill utilization will be assessed via a daily in-app checklist for patients (including an option to report "none").

OTHER OUTCOMES:
Change in Therapist Treatment Fidelity | Weekly during the 12-week intervention period
  The investigators will adapt clinician-rated checklists adapted from past research to identify which components of the Unified Protocol were used by therapists as a treatment fidelity check.
Clinical Utility | 12-week
  The investigators will administer the Clinical Utility Rating Form (CURF), to assess utility of STAR. Questions ask about utility of assessment information and modules for formulating a treatment plan, anticipating treatment difficulties, clinical communication, etc.
Discharge Decisions | 12-week
  At baseline and end-of-treatment, clinicians will be asked to provide information about their discharge decision (e.g., transition to higher or lower level-of-care, discontinuation due to improvement, and discontinuation against medical advice). From randomization until discharge or end of 12-week period, whichever is first.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsie Forbush, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Wakarusa Research Facility, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected from this study will be made publicly available. The investigators will restrict any data that may reveal subjects' identities (e.g., geographical location). To protect subjects' privacy, publicly-available data will not contain any personally identifying or private health information (PHI). Consent forms will describe the data sharing plan so that participants are informed of how their data will be handled. Prior to the release of data, the investigators will require that a local privacy officer certify that all datasets contain no PHI. The investigators will also require that individuals requesting data sign a Letter of Agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be released in a timely fashion in waves as soon as the main study findings are published. Data will remain available in perpetuity.
Access Criteria: Investigators interested in using the data will be required to contact the PI to provide a brief description of the intended use. Although investigators will be able to design and analyze the data as they choose, such documentation will prevent duplication of research and provide a greater level of protection of intellectual property. These instructions will be included in a peer-reviewed publication that describes the study design.